CLINICAL TRIAL: NCT05402189
Title: Ketodex Versus Opioid Based Anaesthesia in Cleft Palate Repair
Brief Title: Ketodex Versus Opioid Based Anaesthesia in Cleft Palate Repair Ketodex Versus Opioid Based Anaesthesia in Cleft Palate Repair Ketodex Versus Opioid Based Anaesthesia in Cleft Palate Repair Ketodex Versus Opioids in Cleft Palate Repaire
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Marwa Emam, Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU R 10 2022
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Ketodex Versus Opioids Based Anaesthesia in Cleft Palate Repair
Keywords: Ketodex, opioids, cleft palate
MeSH Terms: conditions — Cleft Palate | interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: prospective interventional randomized study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed using a computer-generated random number table in opaque sealed envelopes with 1:1 allocation ratio by an anesthesiologist not directly involved in the trial or patient care.
  - Patients will be subsequently followed up by a researcher who will be unaware of the group allocation. Thus effectively, the patient and the outcome assessor will be blinded to the group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketodex group : Group (KD) (Active Comparator)
  Interventions: Drug: Ketodex, Fentanyl
- Opioid group: Group (OP) (Active Comparator)
  Interventions: Drug: Ketodex, Fentanyl

INTERVENTIONS:
Drug: Ketodex, Fentanyl — The patients will be randomized into 2 groups : group (KD) and group (OP) . Two 20 ml syringes, labelled loading and another two 20 ml syringes labelled maintenance will be given to each patient according to his group.
  Group (KD): patients will receive 1mg/kg ketamine and 1ug/kg dexmiditomidine in their respective loading syringes diluted in 20ml normal saline. Then , they will receive ketamine 0.1 mg/kg /hr and dexmedetomidine0.2ug/kg/hr in their maintenance syringes prepared in 20 ml normal saline in a concentration of 1mg/ml ketamine and 1ug/ml dexmiditomidine respectively .
  Group (OP): one of the loading syringes will contain fentanyl in a dose of 2ug/kg diluted in 20 ml normal saline and the other loading syringe will contain normal saline. Then, the patients will receive 0.5ug/kg/hr fentanyl through one of the maintenance syringes while the other syringe contains normal saline.

SUMMARY:
This study will be conducted to compare Ketodex versus opioid based anaesthesia in cleft palate repair surgeries .

DETAILED DESCRIPTION:
According to patients' randomized groups, study medication is given at induction and continues intraoperative not more than 2hours.[8]. Induction of anaesthesia with inhalational anaesthetic will be done through a face mask and Ayres T piece (sevoflurane )8%on 100% oxygen and fresh gas flow of at least double patient minute volume and IV line will be inserted and secured in place .After confirmation of intermittent positive pressure ventilation , 1.5 mg/kg IV suxamethonium will injected. The child will be intubated with an appropriate sized tube, and a throat pack will be placed. Ventilation will be performed with a standard ventilator equipped with a paediatric circle circuit (Datex Ohmeda, Helsinki, Finland), tidal volume of 6-8 ml/kg, and a rate adjusted to maintain the ETCO2 concentration between 32 and 35 mmHg at a total gas flow of 2 L/min. General anaesthesia will be maintained with 50% O2 + 50% air with atracurium and isoflurane, which will be titrated according to the hemodynamic parameters. Dexamethasone (0.2 mg/kg) will be given as an antiemetic and to reduce airway oedema. Post-intubation, Group (KD) will receive 1mg/kg IV ketamine and 1 µg/kg dexmiditomidine IV diluted in 20 ml NS as a loading dose over 10 min followed by a maintenance infusion of ketamine at 0.1 mg/kg/hr and dexmiditomidine 0.2 µg/kg/hr. IV diluted in 20 ml NS till the end of surgery.(15-16-17) Group (OP) will receive fentanyl 2ug /kg IV diluted in 20 ml NS and another loading syringe containing 20 ml normal saline as a loading dose over 10 min followed by a maintenance infusion of another 20 ml syringes, one containing fentanyl and the other containing normal saline . Maintenance dose of fentanyl in this group will be 0.5 µg /kg/hr . Pre-operative fasting fluid deficits and intraoperative losses will be replaced with crystalloid. A single shot of intravenous antibiotic will be given. At the end of surgery, patients will be reversed with 0.05mg/kg IV neostigmine and 0.02 mg/kg atropine, and extubated after meeting the standard extubation criteria

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 5 years; both sex, American Society of anaesthesiologists' physical status I or II; no associated any other congenital anomalies.

Exclusion Criteria:

* Patients with a history of prematurity delayed motor , mental or developmental milestones, long QT syndrome, are excluded from the study allergy to study drugs

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
postoperative respiratory depression | 4 months after starting the study
  This study will be conducted to compare Ketodex versus opioid based anaesthesia in cleft palate repair surgeries as regard postoperative respiratory depression and the need for oxygen

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt